CLINICAL TRIAL: NCT05598931
Title: Development of Neuro-Navigated Transcranial Magnetic Stimulation (TMS) Using MRI
Status: Completed | Type: Observational
Sponsor: Soterix Medical (Industry)
Collaborators: Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: SMICU061621B
Record Dates: First submitted 2021-06-16; First posted 2022-10-28 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Healthy Controls: Subjects will undergo a single MRI session and will then participate in an on-line neuro-navigation session in which various TMS coil positions will be recorded. The brain/head images will be provided to the programmer to permit development of the virtual neuro-navigation algorithm. Data from Yr1 will be used by the programmer as a training sample, and from Yr2 as a test sample.
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — Subjects will participate in an on-line neuro-navigation session in which 6 TMS coil positions will be recorded.

SUMMARY:
Healthy controls (HC) will be studied once to provide data needed to validate the virtual neuro-navigation system. All subjects will undergo a single MRI session and will then participate in an on-line neuro-navigation session in which various TMS coil positions will be recorded. The brain/head images will be provided to the programmer to permit development of the virtual neuro-navigation algorithm. Data from Yr1 will be used by the programmer as a training sample, and from Yr2 as a test sample.

DETAILED DESCRIPTION:
HC subjects (n=10)/yr will be studied once to provide data needed to validate the virtual neuro-navigation system. All subjects will undergo a single Human Connectome Project compatible MRI session permitting application of both surface-based and more standard volumetric analyses. Subjects will then participate in an on-line neuro-navigation session in which TMS coil positions (in 10/20 coordinate space) will be recorded corresponding to the following targets: 1) hand-representation of motor strip; 2) 5-cm location; 3) 5.5 cm location; 4) MNI coordinates corresponding to the "Fitzgerald"4 and "Weigand"6 volumetric targets; 5) peak anti-correlated region (calculated from rsfcfMRI data alone); 6) center of our targeted parcel, calculated using surface-based approaches. The brain/head images will be provided to the programmer to permit development of the virtual neuro-navigation algorithm. Data from Yr1 will be used by the programmer as a training sample, and from Yr2 as a test sample. The Go/No-go criterion is an interclass correlation coefficient (ICC) of >.9 between scalp coordinates determined by on-line neuro-navigation and those determined virtually

ELIGIBILITY:
Inclusion Criteria:

* Non-depressed subjects

Exclusion Criteria:

* Ever met criteria for a psychotic disorder (Sz, SzAff, Bipolar disorder); anorexia nervosa or bulimia nervosa within the last year
* Unstable medical condition by history, physical exam or laboratory results
* Contraindications to MRI (based on metal screening form)
* Meets criteria for claustrophobia
* Recent drug or alcohol use disorder with DSM-5 specifier of moderate or severe within 6 months, or mild within 2 months; lifetime history of IV drug use
* A neurological or neuromuscular disorder;
* Require medications for a general medical condition that contraindicate the TMS treatment
* History of ketamine treatment within 6 mo
* History of monoamine oxidase inhibitor (MAOI) within the past month
* Lacks capacity to consent
* Taking medications that increase the risk of seizures. For patients on permitted concomitant psychotropic agents (antidepressants, anticonvulsants, benzodiazepines, hypnotics, opiates, triiodothyronine (T3), modafinil, psychostimulants, buspirone, melatonin, omega-3 fatty acids, folate, lmethylfolate, s-adenosyl methionine, lithium) dosing must be stable for at least four weeks prior to study entry

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Healthy Controls
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Brain Coordinates | Day 1
  MRI based brain coordinates will be determined using newly developed neuronavigation software

CONTACTS AND LOCATIONS:
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No